CLINICAL TRIAL: NCT04484376
Title: Predictive Factors of Mortality in Invasive Fungal Disease in Post-surgical Critical Care Unit
Acronym: FPR-IIS
Status: Completed | Type: Observational
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Principal Investigator, Hospital Universitario La Fe
Other Study IDs: FPR-IIS -029-02 Ed. 03
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Fungal Invasive Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Other invasive candida infection: Patients with invasive candida infection due a Candida specie othr than Candida Auris.
- Candida Auris related invasive infection: Candida Auris related invasive candida infection.

SUMMARY:
Invasive fungal disease in the critically ill patient is a serious complication that increases hospitalization times, morbidity and mortality, and healthcare costs.

Our team proposes a retrospective observational study of patients from the resuscitation unit of the Hospital la Fe who during the years 2016-2019 presented invasive candidiasis. The investigators intend to detect if there are possible specific risk factors that favor the development of invasive candidiasis in colonized patients and if these associated risk factors could be considered as 'triggers' or alerts for the implementation of specific care in these patients.

To do this, the investigators intend to study the blood samples taken from patients, taking into account different types of perioperative variables from them, which will be statistically analyzed, so that evidence-based inferences can be drawn to demonstrate our hypothesis.

DETAILED DESCRIPTION:
The hypothesis is that there are factors predisposing to the development of invasive fungal disease, invasive candidiasis, and that the detection of these factors may allow detecting the population at risk and implementing both pharmacological measures and general strategies to reduce the mortality of fungal infection.

Primary objective: To determine if candida auris is associated with increased risk of mortality in invasive fungal disease and the risk factors for mortality in the invasive fungal disease, including the species of candida that causes this disease.

Secondary objectives:

Determination of predictors of mortality in invasive fungal disease. Prepare and validate a score in our environment that allows discriminating those patients with a high risk of mortality.

To analyze the pharmacological management that has been carried out in patients who develop candidemia due to auris.

Detect hospital stays of both population groups, in terms of health management.

Type of study: observational, longitudinal, and retrospective study of cases and controls of a selected exposed population that developed the disease over time or not.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years
* Admitted to the ICU that present fungal invasive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population included in the study will be adult patients over 18 years admitted to the Reanimation unit who present fungal invasive disease during their admission to the unit in the period between May 2016 and January 2019.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Patients mortality | Hospital stay (up to 6 months)
  Number of patients with fungal disease related fatal outcome from diagnosis to end of hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital la Fe, Valencia, Spain